CLINICAL TRIAL: NCT05749146
Title: Palliative Care at Home for Patients With Dementia and Their Caregivers
Brief Title: Palliative Care for Patients With Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Laura Gelfman, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: GCO 19-1232; R01AG067045 (NIH)
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: Subjects assigned to intervention or control arms in a 1:1 ratio
Who Masked: Outcomes Assessor
Masking Description: Single blind control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palliative care at home (Experimental): Randomized to intervention arm
  Interventions: Behavioral: Home Palliative Care
- Augmented control (Active Comparator): Randomized to augmented control (visits to the caregiver from a CHW without training in dementia or palliative care)
  Interventions: Behavioral: Home Palliative Care

INTERVENTIONS:
Behavioral: Home Palliative Care — Patients/caregivers will be cared for by an interdisciplinary team that includes a social worker, nurse, community health worker, nurse practitioner, and physician.

SUMMARY:
A multi-site, single-blinded, parallel, randomized-controlled trial to evaluate the effectiveness of a novel model of in-home palliative care for dementia patients and their family caregivers. From inpatient and outpatient settings associated with four hospitals across New York City, patients with advanced dementia and their family caregivers will be randomized to intervention or augmented control.

DETAILED DESCRIPTION:
The objective of this randomized controlled trial is to study the impact of a new home based palliative care program on patients' symptoms, quality of life, satisfaction with care, completion of advance care planning documentation and receipt of care consistent with preferences. In addition, the study will examine the impact of this model of care on patient healthcare utilization, including hospitalization, emergency department utilization, and hospice use prior to death. The trial will also include patients' caregivers, in order to examine the impact of the intervention on caregiver burden and prevalence of depression.

Patients randomized to the intervention will be scheduled for an intake visit. This visit will be undertaken by the team's registered nurse and/or social worker, together with a community health worker, and other team members (advanced practice nurse, MD), depending on patients' needs. Visits will combine a combination of video-teleconferencing technology and in person visits. Following this visit, and in conjunction with the nurse practitioner and/or MD, a care plan will be developed to address areas of clinical need highlighted during the intake visit.

Patients in the intervention arm will receive ongoing monitoring and input (telephone-based, video-based, and in-person) from members of the clinical team, dependent on their identified needs. Patients' cases will be discussed at the weekly IDT meeting, as appropriate to the level of clinical need. Patients and caregivers will be provided with access to a 24 hour telephone line, staffed by a Mount Sinai based physician, which acts as an advice line out of hours. These physicians will be able to provide advice to patients and caregivers.

ELIGIBILITY:
Inclusion Criteria:

* have advanced dementia, based on Global Deterioration Score (GDS)>6
* impairment in at least one activity of daily living (ADL -which is inherent in this level of GDS)
* at least one hospitalization or ED visit within the last 12 months
* a physician who is primarily responsible for their dementia-related care whose clinical outpatient site is associated with one of the four Mount Sinai sites in Manhattan
* a family caregiver willing to enroll
* a residence in Manhattan where they are currently living (not in a long-term care facility)
* capacity to consent or a legal representative available to provide consent
* fluency in English or Spanish, or their legal representative must be fluent in English or Spanish
* age >64.

Exclusion Criteria:

* Does not have a family caregiver to enroll
* Does not reside in Manhattan outside of long-term care facility
* Does not have fluency in English or Spanish Doesn't

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Symptom Management as measured by the End of Life for Dementia scale | 6 months
  This will be determined using a validated structured questionnaire administered to patient-subjects or caregiver via telephone interview or in person by the trained research coordinator. The Symptom Management at the End of Life in Dementia (SM-EOLD) scale responses range from 0 to 45 with higher scores indicating better symptom management.

SECONDARY OUTCOMES:
Number of Hospital Admissions | at 12 months
  Acute care utilization as measured by the number of hospital admissions
Number of Hospital Stays | at 12 months
  Acute care utilization as measured by the number of hospital days
Patient reported treatment concordance | at 12 months
  The Study Team will examine if the care patients receive is concordant with the care they wanted to receive using simple chart review of whether care received matches stated preferences (yes/no).
Cost Analysis | at 12 months
  Total costs between the arms including inpatient, emergency department, ambulatory services, and home care services will be compared. Costs of the clinical intervention (e.g. clinical personnel, transportation) will be included in the analyses.
Caregiver burden per Zarit Burden Inventory | at 6 months
  Zarit Burden Inventory to determine caregiver burden by using a validated structured 22-item questionnaire administered to caregiver-subjects via telephone interview or in person by the trained research coordinator. Each item is on a 5-point scale range from 0 (never) to 4 (always). Full scale from 22 - 110, higher score indicates a greater burden.
Caregiver burden per Zarit Burden Inventory | at 12 months
  Zarit Burden Inventory to determine caregiver burden by using a validated structured 22-item questionnaire administered to caregiver-subjects via telephone interview or in person by the trained research coordinator. Each item is on a 5-point scale range from 0 (never) to 4 (always). Full scale from 22 - 110, higher score indicates a greater burden.
Caregiver satisfaction measured using FAMCARE-10 | at 6 months
  FAMCARE-10 to assess caregiver satisfaction by using a validated 10-item structured questionnaire administered to patient-subjects via telephone interview or in person by the trained research coordinator. Full scale ranges 0-20, with higher scores indicating higher satisfaction.
Caregiver satisfaction measured using FAMCARE-10 | at 12 months
  FAMCARE-10 to assess caregiver satisfaction by using a validated 10-item structured questionnaire administered to patient-subjects via telephone interview or in person by the trained research coordinator. Full scale ranges 0-20, with higher scores indicating higher satisfaction.
Caregiver depression measured by PHQ-9 Score | at 6 months
  PHQ-9 to assess Caregiver Depression by using a validated structured 9 item questionnaire administered to caregiver-subjects via telephone interview or in person by the trained research coordinator. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Full scale from 0-27, with higher score indicating more severe symptoms.
Caregiver depression measured by PHQ-9 Score | at 12 months
  PHQ-9 to assess Caregiver Depression by using a validated structured 9 item questionnaire administered to caregiver-subjects via telephone interview or in person by the trained research coordinator. The PHQ-9 is the depression module, which scores each of the 9 DSM-IV criteria as "0" (not at all) to "3" (nearly every day). Full scale from 0-27, with higher score indicating more severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Laura P Gelfman, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Ichan School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  For individual participant data meta-analysis. Proposals should be directed to christian.espino@mssm.edu. To gain access, data requestors will need to sign a data access agreement.